CLINICAL TRIAL: NCT01902394
Title: The Addition of Whole Grains to the Diets of Adults: A Study of Digestive Health and Natural Defenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: General Mills (Industry); Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Simin Meydani, Director of the Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2720
Record Dates: First submitted 2012-06-04; First posted 2013-07-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Digestive Health and Immune Function
Keywords: digestive health and natural defenses
MeSH Terms: interventions — Whole Grains

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole grain rich diet (Experimental): Participants in the whole grain (WG) group will receive a diet providing 100% of energy requirements in a diet rich in whole grains.
  Interventions: Other: Whole grains
- Refined grain rich diet (Placebo Comparator): Participants in the refined grain (RG) group will receive a diet providing 100% of energy requirements in a diet rich in refined grains.
  Interventions: Other: Refined grains
- Negative control (No Intervention): Subjects randomized to the negative control group will consume their own usual diet (i.e. not receive foods and beverages from the study).

INTERVENTIONS:
Other: Whole grains — Following completion of the baseline period (a 2-week run-in phase), participants in the WG group will receive a diet providing 100% of energy requirements in a diet rich in whole grains and the RG group will be provided with 100% of energy requirements in a diet rich in refined grains but otherwise similar to the WG diet for 6 weeks.
  Arms: Whole grain rich diet
Other: Refined grains — Following completion of the baseline period (a 2-week run-in phase), participants in the WG group will receive a diet providing 100% of energy requirements in a diet rich in whole grains and the RG group will be provided with 100% of energy requirements in a diet rich in refined grains but otherwise similar to the WG diet for 6 weeks.
  Arms: Refined grain rich diet

SUMMARY:
The purpose of this study is to determine if substituting whole grains for refined grains in the diets of healthy adults over a period of 6 weeks alters the composition of the bacteria in the gut, and has beneficial effects on immune function, digestive health, cardiovascular health, regulation of body weight and composition, and vitamin K status.

The investigators hypothesize that whole grain consumption over a period of 6 weeks will alter the gut microflora toward a more beneficial bacterial profile, improve the immune response while reducing oxidative stress and inflammatory markers, have favorable effects on factors influencing the regulation of body weight and composition,increase bacterial vitamin K synthesis, and beneficially effect surrogate markers of cholesterol synthesis/absorption, vitamin D concentrations, and whole genome DNA methylation patterns. In statin users it is hypothesized that, consumption of whole grains will alter statin pharmacokinetics by decreasing rate of statin absorption, resulting in more sustained plasma concentrations.

DETAILED DESCRIPTION:
This study is a randomized parallel-arm trial using a six-week dietary intervention following a 2 week run-in period. Healthy volunteers will be randomized to two groups (n=40/group), and consume either a diet rich in whole grains or a diet rich in refined grains provided at estimated energy requirements for 6 weeks. Outcomes will be measured during the run-in period and at week 6 of the intervention. To control for variation in microbiota an additional 10 volunteers will serve as "negative controls" and not undergo any diet intervention.

ELIGIBILITY:
Subjects Inclusion Criteria

* Healthy male and female subjects aged 40-65 y (women must be > 1 year postmenopausal or had both ovaries removed, if premenopausal).
* Body mass index (BMI) 20-35 kg/m.2
* Pass screening blood and urine tests

  * Creatinine ≤ 1.5 mg/dL
  * glutamic oxaloacetic transaminase/serum glutamate pyruvate transaminase/total bilirubin ≤ twice the upper limit of normal range
  * Fasting glucose <125 mg/dL
  * hematocrit ≥ 32%
  * white blood cell count ≥ 1.8 x 103/mm3 (M)
  * PLT ≥ 100 x 103/mm3 (thou/µL)
* Must be willing to be randomized.
* Those randomized to either the WG or RG groups must be willing to consume only study foods and beverages provided.

Exclusion Criteria

* Self reported weight change >4kg within the past 3 months.
* Have participated in a weight loss program within the last 3-months; eligible if in weight reduction program to maintain body weight.
* Not willing to reduce habitual daily fiber intake (including prebiotics) within 2 wk prior to enrollment to < ~7g/1000kcal/d for men, or <~8g/1000kcal/d for women if currently consuming greater amounts.
* Not willing to stop consumption of probiotic or prebiotic supplements within 2 weeks prior to start of study if currently taking these, as well as during study participation.
* Vegetarian diet.
* Not willing to stop taking multivitamins, and supplements (with the exception of vitamin D and calcium), including fish oil or n-3 fatty acids and herbal supplements, for 30 days prior to or during study participation, if currently taking these.
* Regular use of laxatives, stool softeners, or anti-diarrheal medications, and medications influencing food intake and/or appetite.
* Not willing to undergo a 3-month washout period after colonoscopy prior to enrollment, and not willing to defer colonoscopy until after study completion.
* Eating disorder within the past 10 years.
* Disinhibited eating behavior as indicated by a score above 12 on the Three Factor Eating Questionnaire.
* Food allergies or aversions or other issues with foods that would preclude use of study diets, including gluten, milk, nuts, or eggs.
* Individuals identified during screening as having barriers expected to deter compliance with dietary requirements (e.g., stated dislike of study foods, inadequate resources to store and reheat meals, inability to adhere to food pick-up schedule).
* Alcohol consumption >2 drinks per day.
* Not willing to abstain from alcohol consumption during the study.
* Smoking or using nicotine containing products in the last 6 months.
* Use of aspirin, non-steroidal anti-inflammatory medications (NSAIDs) or antihistamine prescribed by a physician or clinician, or the inability to discontinue the use of these substances for 72 hrs before first day blood draw until 48 hrs after DTH implant (i.e. after second reading).
* Use of anabolic steroids, insulin, growth hormone or testosterone.
* Type I or type II diabetes.
* Uncontrolled major illnesses. (Will include if stable on drugs used to control cardiovascular, liver, and renal diseases, asthma, and dysphagia).
* Current use of proton pump inhibitors and H2 blockers to control acid-reflux/heart burn
* Use of medications which interfere with energy metabolism including oral glycemic agents and insulin.
* Uncontrolled hypertension as determined by study physician or nurse.
* Use of immunosuppressive drugs.
* Active cancer or current cancer diagnosis (except non-melanoma skin cancer).
* Active infection within 2 weeks of study enrollment, blood draws or skin tests; however, may participate if admission is postponed or study activity is rescheduled > 2 weeks after resolution of symptoms.
* Any antibiotic use within the past 3 months, except topical antibiotic use.
* History of dysphagia, malabsorptive disorders, inflammatory bowel disease or other gastrointestinal disorders such as ulcerative colitis, Crohn's disease, celiac disease , chronic diarrhea or constipation.
* Gastric bypass or other surgery for weight loss.
* Splenectomy or partial splenectomy.
* Autoimmune diseases such as rheumatoid arthritis and psoriasis. Autoimmune thyroid disease that has been treated and with stable replacement doses is not an exclusion.
* Taking warfarin or coumadin any time during the previous 6 months.
* Current diagnosis of or treatment for psychosis (i.e. schizophrenia, etc.). Include depression if has been stable on treatment regimen for > 6 months.
* Blindness or deafness not corrected with use of glasses and hearing aids.
* Does not speak English; due to insufficient funds to hire a translator and to get all study materials translated into another language to allow us to recruit non-English speaking participants non-English speakers will not be eligible to participate.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in T Cell-mediated immunity | week 2 of washout diet and week 6 of diet intervention
  Delayed-type hypersensitivity (DTH) and lymphocyte proliferation will be measured at baseline (week 2 of washout period) and at week-6 of the diet intervention to assess adaptive immune function, specifically T cell-mediated immunity.
change in Lymphocyte proliferation | week 2 of washout diet and week 6 of diet intervention
  Whole blood collected at baseline (week 2 of washout period) and at week-6 of the diet intervention will be investigated for the ability of lymphocytes to proliferate by quantifying the incorporation of tritium following mitogen stimulation.
change in Natural Killer Function | week 2 of washout diet and week 6 of diet intervention
  The ability of peripheral blood mononuclear cells to bind and kill leukemia cells will be measured at baseline (week 2 of washout period) and at week-6 of the diet intervention
change in Cytokines | week 2 of washout diet and week 6 of diet intervention
  Peripheral blood and stool samples will be analyzed at baseline (week 2 of washout diet) and week-6 of diet intervention for cytokines.
change in Salivary immunoglobulin A (IgA) | week 2 of washout diet and week 6 of intervention diet
  Salivary IgA will be analyzed at baseline (week 2 of washout period) and at week-6 of the diet intervention.

SECONDARY OUTCOMES:
change in gut microbiota composition | week 2 of washout diet and week 6 of intervention diet
  Phylogenetic composition and relative abundance of bacteria in stool will be analyzed from 24-hour fresh sample collected at baseline (week 2 of washout diet) and at week 6 of intervention diet
change in cardiovascular health risk factors | week 2 of washout diet and week 6 of intervention diet
  Consumption of the whole grain (WG) diet will be beneficial for multiple outcomes of cardiovascular health including a favorable blood lipid profile (low density lipoprotein, very low-density lipoprotein, high density lipoprotein, total cholesterol and triglycerides), and a decrease in blood pressure, and in oxidative stress status (secondary hypothesis).
change in vitamin K status | week 2 of washout diet and week 6 of intervention diet
  Fecal menaquinones concentrations; Fasting serum phylloquinone and menaquinones concentration from 72-hour stool collected at baseline (week 2 of washout diet) and at week 6 of intervention diet
change in body composition | week 2 of washout diet and week 6 of intervention diet
  Fat and fat free mass; waist and hip circumference
change in appetite | Weekly for 8 weeks
  Visual analog scales to assess hunger, fullness and satisfaction while on the study diet
change in fasting gut hormone concentration | week 2 of washout diet and week 6 of intervention diet
  Plasma glucagon-like peptide-1 and peptide-YY will be measured from blood samples collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in fasting serum leptin | week 2 of washout diet and week 6 of intervention diet
change in glycemic regulation | week 2 of washout diet and week 6 of intervention diet
  48 hr continuous glucose monitoring; fasting serum glucose; fasting serum insulin; HOMA-IR
change in resting energy metabolism | week 2 of washout diet and week 6 of intervention diet
  Resting energy expenditure; substrate oxidation at rest
change in eating behaviors | week 2 of washout diet and week 6 of intervention diet
  Questionnaires will be administered at baseline (week 2 of washout diet) and week 6 of intervention diet
change in quality of life | week 2 of washout diet and week 6 of intervention diet
  Questionnaires will be administered at baseline (week 2 of washout diet) and week 6 of intervention diet
change in breath hydrogen and methane | week 2 of washout diet and week 6 of intervention diet
change in stool pH | week 2 of washout diet and week 6 of intervention diet
  Will be measured from 72-hour stool sample collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in 72hr fecal weight | week 2 of washout diet and week 6 of intervention diet
  Will be measured from 72-hour stool sample collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in stool water content | week 2 of washout diet and week 6 of intervention diet
  Will be measured from 72-hour stool sample collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in total stool anaerobic and aerobic bacterial counts | week 2 of washout diet and week 6 of intervention diet
  Will be measured from 72-hour stool sample collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in stool energy content | week 2 of washout diet and week 6 of intervention diet
  Will be measured from 72-hour stool sample collected at baseline (week 2 of washout diet) and week 6 of intervention diet
change in DNA methylation | week 2 of washout diet and week 6 of intervention diet
change in concentrations of the cholesterol synthesis (squalene, desmosterol, lathosterol) and absorption (campesterol, sitosterol, cholestanol) markers | week 2 of washout diet and week 6 of intervention diet
  Plasma squalene, desmosterol, lathosterol), campesterol, sitosterol, and cholestanol concentrations will be measured at baseline (week 2 of washout diet) and week 6 of intervention diet
change in serum vitamin D | week 2 of washout diet and week 6 of intervention diet

CONTACTS AND LOCATIONS:
Overall Officials: Simin N Meydani, DVM, PhD, Principal Investigator — Human Nutrition Research Center on Aging; Junaidah B Barnett, MCH(N), PhD, Study Director — Human Nutrition Research Center on Aging
Locations (1):
- HNCRA at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Karl JP, Meydani M, Barnett JB, Vanegas SM, Barger K, Fu X, Goldin B, Kane A, Rasmussen H, Vangay P, Knights D, Jonnalagadda SS, Saltzman E, Roberts SB, Meydani SN, Booth SL. Fecal concentrations of bacterially derived vitamin K forms are associated with gut microbiota composition but not plasma or fecal cytokine concentrations in healthy adults. Am J Clin Nutr. 2017 Oct;106(4):1052-1061. doi: 10.3945/ajcn.117.155424. Epub 2017 Aug 16. PMID 28814395
- [Derived] Vanegas SM, Meydani M, Barnett JB, Goldin B, Kane A, Rasmussen H, Brown C, Vangay P, Knights D, Jonnalagadda S, Koecher K, Karl JP, Thomas M, Dolnikowski G, Li L, Saltzman E, Wu D, Meydani SN. Substituting whole grains for refined grains in a 6-wk randomized trial has a modest effect on gut microbiota and immune and inflammatory markers of healthy adults. Am J Clin Nutr. 2017 Mar;105(3):635-650. doi: 10.3945/ajcn.116.146928. Epub 2017 Feb 8. PMID 28179226
- [Derived] Karl JP, Meydani M, Barnett JB, Vanegas SM, Goldin B, Kane A, Rasmussen H, Saltzman E, Vangay P, Knights D, Chen CO, Das SK, Jonnalagadda SS, Meydani SN, Roberts SB. Substituting whole grains for refined grains in a 6-wk randomized trial favorably affects energy-balance metrics in healthy men and postmenopausal women. Am J Clin Nutr. 2017 Mar;105(3):589-599. doi: 10.3945/ajcn.116.139683. Epub 2017 Feb 8. PMID 28179223